CLINICAL TRIAL: NCT02191943
Title: Long-term Bi-center Trial to Compare the Radiological Cavity Progression of Approximal Caries Following Infiltration or Standard Treatment
Brief Title: Lesion Progression of Approximal Caries After Resin Infiltration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Collaborators: Dep. Conservtive Dentistry, Periodontology and Preventive Dentistry Hannover (Unknown); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CHARM
Record Dates: First submitted 2014-06-20; First posted 2014-07-16 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2014-07

CONDITIONS: Proximal Caries
Keywords: caries; proximal; non-cavitated; fluoridation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (fluoride varnish) (Active Comparator)
  Interventions: Device: Duraphat
- resin infiltration (Icon) (Experimental)
  Interventions: Device: Icon approximal caries infiltration kit

INTERVENTIONS:
Device: Duraphat — The subjects in the control group will be the subject of personalized oral hygiene instructions on the basis of obtained indices, and will also receive a professional prophylaxis. Following this, the surfaces of the teeth in the control group involved in the trial will be treated with a fluoride varnish (Duraphat®) that will be applied with a brush to all surfaces of the teeth, working the varnish approximally with the brush. This treatment will be repeated in the comparative group at each follow-up appointment.
  Other Names: fluoride varnish
  Arms: Control (fluoride varnish)
Device: Icon approximal caries infiltration kit — Carious lesions in the teeth in the test group shall be treated with the infiltrant ICON® according to the manufacturer's instructions. Step by step instructions for application are as follows:
  Other Names: resin infiltration
  Arms: resin infiltration (Icon)

SUMMARY:
The aim of the planned in-vivo trial is to investigate the effectiveness of the caries infiltration technique for the repression of caries progression.

Within the framework of this investigation it is intended that the hypothesis to be substantiated is that carious cavities, which have been treated with the caries infiltration technique, exhibit significantly reduced radiological progression than those cavities that have been treated using standard preventive treatments.

In this multicenter trial, a total of 90 test subjects are included and 45 test subjects at each institution are to be treated with both, the infiltration technique and using conventional fluoridation treatment in different sides of the mouth ("split-mouth design").

The anticipated result of this trial shall deliver information on the long-term effectiveness of caries infiltration to prevent the progression of existing approximal carious lesions, and thereby enable an improvement in caries prevention within the scope of dental treatment.

DETAILED DESCRIPTION:
The aim of the planned in-vivo trial is to investigate the effectiveness of the the caries infiltration technique for the repression of approximal caries progression. .

Within the framework of this investigation it is intended that the hypothesis be substantiated that carious cavities, which have been treated with the caries infiltration technique, exhibit significantly reduced radiological progression than those cavities that have been treated using standard treatments.

Modern dentistry, which is focused more towards preventive and minimally invasive treatment, attempts - with the aid of fluoride therapies and improved oral hygiene - to prevent the onset and progression of carious lesions as much as possible.

Even today, approximal lesions pose a particular problem to the treating dentist. A primary reason for this is the difficulty accessing the localized area of the carious cavity. Treating this area usually requires invasive treatment, in which healthy tooth structure must be removed. Furthermore, it is possible that the filling material may deteriorate as a result of the aging process, meaning that the restoration will require replacement at some point in the future. In order to prevent this, the development of a treatment oriented towards prevention and minimal invasion is key.

For a number of years there has been an option to seal pits and fissures on the occlusal surfaces, which is assessed in the literature as being highly efficacious and effective (Splieth et al. 2010, Ahovuo-Saloranta et al. 2008, Griffin et al. 2008). It constitutes a vital component of the caries prevention approach especially in the event of an increased risk of caries (Hiiri et al. 2010). In recent years there has been an attempt to transfer this treatment concept to applications in the approximal area, in order to prevent unnecessary substance ablation. A fissure sealing resin and a dental adhesive were used for the first time in an attempt at creating a surface diffusion barrier (Gomez et al. 2008, Gomez et al. 2005, Paris et al. 2006, Martignon et al. 2006, Robinson et al. 2001). Coating the tooth surface in the approximal area with various plastic foils after tooth separation opened up a whole new treatment approach for dealing with these carious lesions (Alkilzy et al. 2010, 2009).

The caries infiltration technique constitutes an additional new treatment concept. Here, the surface alone is not exclusively coated but a diffusion barrier is instead created inside the cavity itself, through the penetration of the "infiltrant" into the carious lesion (Paris et al. 2010, Meyer-Lueckel et al. 2010, 2009, 2008, Phark et al. 2009). In current studies, it has been possible to demonstrate inhibition of the progression of carious lesions with the infiltration technique, both in bovine teeth in situ and in artificially generated carious lesions in human teeth in vitro (Paris et al. 2010).

The development of the infiltration technique started back in the 1970's with the first low-viscosity plastic materials. However, these were never put into clinical application due to their toxicity (Robinson et al.1976). During their course of development, adhesive systems were employed for sealing carious lesions (Donly et al. 1992, Garcia-Godoy et al. 1997). These also exhibit a caries-inhibiting effect. However, it has only been possible to determine limited penetration depths. The reason for this is the surface morphology of the carious cavity, with a very limited pore volume on the surface, and the characteristics of the adhesive itself (Paris et al. 2007). In order to facilitate removal of the limiting surface layer, a hydrochloric acid gel was used for the infiltration technique in place of orthophosphoric acid gel for the adhesive technology. Using this conditioner it was possible to guarantee better penetration of the materials up to a depth of 58 µm due to an erosive removal of the surface layer (Meyer-Lueckel et al. 2007, Paris et al. 2007, 2009). In order to better utilize the capillary effect in the altered surface and to thereby increase the penetration depth of the material, monomer mixtures were developed with a high penetration coefficient. These enable a fast penetration of the infiltrant into the altered carious surface up to a depth of 750 µm (Paris et al. 2007, 2009). The sealing of the carious cavity is now no longer restricted to the surface alone, but also encompasses the body of the cavity.

The anticipated result of this trial shall deliver information on the long-term effectiveness of caries infiltration and thereby result in an improvement in caries prevention within the scope of dental treatment, and prevent the progression of existing carious lesions . This is a micro-invasive form of treatment, which largely facilitates the delay or avoidance of conventional invasive initial dental treatment with the associated inevitable loss of healthy tooth structure. Further studies on the optimization of the infiltration technique can be built upon these results. In the long-term, it will be possible to use these findings to develop new prevention and treatment options for approximal carious lesion .

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older
* Good general health
* At least 2 active, approximal caries lesions present without evidence of frank cavitation Caries depth: E2 - D1 (minimum extension to the inner half of the enamel and maximum to the outer third of the dentin)
* The posterior teeth on the upper and lower arches from distal of the first premolar to mesial of the second molar will be included
* All teeth to be treated must have approximal contacts with the adjacent teeth in the arch
* Other teeth requiring treatment will be treated prior to the beginning of the trial
* The patients must declare their consent to participate in the clinical trial following the provision of the required clarifications regarding the method, significance and scope of the trial as well as the associated risks. They may withdraw this consent at any time.
* Participation in the follow-up examinations

Exclusion Criteria:

* - Parallel participation in a further trial relating to dental materials
* The patient has not signed the participant consent form
* Pregnant and breastfeeding women prior to the trial commencing A woman that becomes pregnant after the treatment has been performed will remain in the study, unless she becomes pregnant for a second time in which case, she will be excluded from the study
* Unexplained diseases of the mucous membranes or conditions in the sense of contact allergies to materials used, e.g. oral lichenoid lesions
* Known allergies to ingredients contained within the treatment materials used
* Infectious diseases such as HIV, hepatitis, etc
* Undergoing orthodontic treatment at the time of the trial
* Persons who are presently taking other medication due to other illnesses, which upon our examination are deemed to possibly be a risk or a problem for the patient or the study
* A large number of existing carious lesions that have not been restored and would require extensive treatment, comprehensive prosthetic restorations that need to be done or replaced and severe periodontal disease
* Current use of bleaching products or use within the two weeks previous to the start of the study
* No assured dry isolation possible as required per the criteria of the adhesive technology (rubber dam system)
* Persons with a history of allergies
* Patients with dental treatment phobias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
progression of non-cavitated proximal caries lesions | up to 36 months
  preventing the progression of non-cavitated approximal lesions in comparison to conventional non invasive treatment; lesion progression will be monitored by annual bitewings and comparison to baseline lesion size

CONTACTS AND LOCATIONS:
Overall Officials: Silke Jacker-Guhr, Dr., Principal Investigator — Department of Conservtive Dentistry, Periodontology and PreventiveDentistry Hannover Medical School; Anne-Kathrin Lührs, Dr., Principal Investigator — Department of Conservtive Dentistry, Periodontology and PreventiveDentistry Hannover Medical School; Jack L Ferracane, Prof., Study Chair — OHSU School of Dentistry / Department of Restorative Dentistry Oregon Health and Science University (OHSU)
Locations (1):
- OHSU School of Dentistry / Department of Restorative Dentistry Oregon Health and Science University (OHSU), Portland, Oregon, United States